CLINICAL TRIAL: NCT06238141
Title: Effects of Expressive Writing on Stress and Work-Related Outcomes Among Student Nurse Interns: a Randomized Controlled Trial
Brief Title: Expressive Writing on Stress and Work-Related Outcomes Among Student Nurse Interns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changzhi Medical College (Other)
Responsible Party: Principal Investigator, JI XUAN, Lecturer, Changzhi Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RT2023047
Record Dates: First submitted 2024-01-24; First posted 2024-02-02 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Stress, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This study is single-blinded. The intervention trainer will not be blinded because a single researcher conducts the study. In order to minimize experimenter bias, outcome assessments will be conducted through an online questionnaire survey platform (Wenjuanxing), with the trainer distributing the same link to all participants. During data collection, only acronyms of the questionnaires will be used to avoid self-fulfilling expectations.
  Participants will be informed during the recruitment phase that the study aims to explore the effect of writing on the internship experience and feelings only. Assignment to the intervention or control group will remain undisclosed to participants until the end of the 3-month follow-up. Participants could unblind themselves by exiting the study and requesting debrief information.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Other: Expressive writing
- control group (Sham Comparator)
  Interventions: Other: Neutral writing

INTERVENTIONS:
Other: Expressive writing — According to the writing prompts, online expressive writing focuses on stressful events and will be conducted twice a week (every Monday and Thursday) for 15 minutes each time, lasting for ten weeks.
  Writing prompts are developed based on Emotional Processing Theory (EPT) and Cognitive Adaptation Theory (CAT).
  Arms: intervention group
Other: Neutral writing — According to the writing prompts, online neutral writing focuses on immediate surroundings and will be conducted twice a week (every Monday and Thursday) for 15 minutes each time, lasting for ten weeks.
  Arms: control group

SUMMARY:
The goal of this interventional study is to assess the effects of an intervention on stress and work-related outcomes among Chinese student nurse interns. The main questions it aims to answer are:

* Does expressive writing reduce clinical practice stress and improve coping strategies in student nurse interns?
* Does expressive writing increase work engagement and perceived professional benefit among student nurse interns?

Participants in the intervention group and control group will perform expressive writing and neutral writing, respectively, based on different given instructions. In both groups, writing will last for 15 minutes each time, twice a week, for ten weeks.

Researchers will compare the outcomes of the two groups to see if there are differences between clinical practice stress, coping strategies, work engagement, and perceived professional benefit.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate student nurse interns in their first clinical internship (had no prior clinical practice experience)
* Have access to and proficiency in utilizing social media
* Be able to read and write via the internet
* Be willing to fill in questionnaires and write according to the assigned writing prompts
* Never participated in expressive writing or stress management intervention programs

Exclusion Criteria:

* Intern at a self-contacted hospital
* Severe current psychological conditions
* Undergoing any form of psychotherapy
* With a habit of keeping diaries

Withdrawal criteria:

* Termination of internship for whatever reason
* Not submit writing materials twice

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-10-27 (Actual); Study Completion 2024-10-27 (Actual)

PRIMARY OUTCOMES:
Mean Change from Baseline in Clinical Practice Stress Scores on the Stress Rating Scale for Nursing Students in Practice at 10 Weeks, 14 Weeks and 18 Weeks | At baseline, post-intervention at Week 10, 14-week, 18-week and 22-week follow-up.
  The scale consists of 6 dimensions and 37 entries, including the nature of work, workload, preparation for an internship, interpersonal relationships, work support, and learning and work impulse. The scale rates on a 4-point Likert scale, with no stress, mild stress, moderate stress, and severe stress, assigned a score of 0, 1, 2, and 3, respectively, and the higher the score, the greater the stress.

SECONDARY OUTCOMES:
Mean Change from Baseline in Positive and Negative Coping Style Scores on the Brief Coping Style Scale at 10 Weeks, 14 Weeks and 18 Weeks | At baseline, post-intervention at Week 10, 14-week, 18-week and 22-week follow-up.
  The scale consists of two dimensions, positive and negative coping, with 20 entries. A 4-point Likert scale is used, with 1-4 indicating "not used" to "often used". Positive coping has 12 entries, and negative coping has 8 entries, with higher scores indicating more frequent use of coping strategies.
Mean Change from Baseline in Work Engagement Scores on the Utrecht Work Engagement Scale at 10 Weeks, 14 Weeks and 18 Weeks | At baseline, post-intervention at Week 10, 14-week, 18-week and 22-week follow-up.
  The scale consists of 3 dimensions: vitality, dedication, and concentration, comprising 15 entries. A 7-point Likert scale is used, with scores ranging from 0-6 for "never," "almost never," "rarely," "sometimes," "often," "frequently," and "always." The total score is the sum of the scores of each entry. An average entry score of 4 or more is defined as a high level of work engagement, 2-4 as a moderate level, and less than 2 as a low level of work engagement.
Mean Change from Baseline in Perceived Professional Benefits Scores on the Perceived Professional Benefits Scale at 10 Weeks, 14 Weeks and 18 Weeks | At baseline, post-intervention at Week 10, 14-week, 18-week and 22-week follow-up.
  The scale consists of 7 items of positive career sense, 6 items of good nurse-patient relationship, 6 items of sense of belonging to the team, 8 items of self-growth, and 6 items of identification with friends and relatives, totaling 33 items in 5 dimensions, and each item is scored 1 to 5 on a 5-point Likert scale ranging from "strongly disagree" to "strongly agree. The higher the score, the stronger the perceived professional benefit.

CONTACTS AND LOCATIONS:
Overall Officials: XUAN JI, Principal Investigator — Changzhi Medical College
Locations (1):
- Changzhi Medical College, Changzhi, Shanxi, China

IPD SHARING:
Plan to Share IPD: Yes
Available by contacting the central contact person after completion of the trial.
Time Frame: from April 2025 to September 2025
Access Criteria: Any reason that can tap into the potential higher value of the data.

DOCUMENTS (2):
  • Study Protocol (2023-10-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT06238141/Prot_000.pdf
  • Informed Consent Form (2023-10-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT06238141/ICF_001.pdf